CLINICAL TRIAL: NCT02061787
Title: the Application of Cardiopulmonary Exercise Testing in Assessment Outcome of Patients With Pulmonary Hypertension
Acronym: CPETPH
Status: Recruiting | Type: Observational
Sponsor: Chinese Pulmonary Vascular Disease Research Group (Other)
Responsible Party: Sponsor
Other Study IDs: CPETPH
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2022-07

CONDITIONS: Pulmonary Hypertension; Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Arterial Hypertension Associated With Schistosomiasis (Disorder)
Keywords: Chronic Thromboembolic Pulmonary Hypertension; Pulmonary Arterial Hypertension; balloon pulmonary angioplasty; cardiopulmonary exercise test
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- cardiopulmonary exercise testing: patients diagnosed with pulmonary hypertension, including pulmonary arterial hypertension or chronic thromboembolic pulmonary hypertension, were evaluated by cardiopulmonary exercise testing before and after medical or balloon pulmonary angioplasty treatment
  Interventions: Device: balloon pulmonary angioplasty

INTERVENTIONS:
Device: balloon pulmonary angioplasty — patients with chronic thromboembolic pulmonary hypertension who underwent balloon pulmonary angioplasty

SUMMARY:
cardiopulmonary exercise test evaluate patients with pulmonary hypertension before and after medical or balloon pulmonary angioplasty treatment

DETAILED DESCRIPTION:
patients diagnosed with pulmonary hypertension, including pulmonary arterial hypertension and chronic thromboembolic pulmonary hypertension, will be evaluated by cardio pulmonary exercise test before and after medical or balloon pulmonary angioplasty treatment

ELIGIBILITY:
Inclusion Criteria:

* pulmonary arterial hypertension;( WHO1)
* chronic thromboembolic pulmonary hypertension;
* pulmonary arterial hypertension due to other cause;

Exclusion Criteria:

* massive hemoptysis;
* unable to accomplish cardiopulmonary exercise testing due to neuromuscular disorders;
* recent recurrent syncope;
* pulmonary hypertension due to hypoxia;
* pulmonary hypertension due to left heart diseases.

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: pulmonary hypertension who may accomplish cardiopulmonary exercise testing.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2010-09 (Actual); Primary Completion 2030-09-08 (Estimated); Study Completion 2030-09-08 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | 5 years
  all cause mortality
mean pulmonary arterial pressure after treatment | 5 years
  the mean pulmonary arterial pressure of patients with chronic thromboembolic pulmonary hypertension after balloon pulmonary angioplasty treatment
achievement of low risk | 5 years
  patients with chronic thromboembolic pulmonary hypertension achievement of low risk after balloon pulmonary angioplasty

SECONDARY OUTCOMES:
deterioration of WHO function | 5 years
  deterioration of WHO function

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, MD，PhD, Study Director — Fuwai Hospital, National Center for Cardiovascular Diseases
Locations (1):
- center of pulmonary vascular disease, Fuwai hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Duan A, Jin Q, Zhang Y, Luo Q, Zhao Q, Yan L, Huang Z, Hu M, Xiong C, Zhao Z, Liu Z. Exercise feature and predictor of prognosis in patients with pulmonary artery stenosis-associated pulmonary hypertension. ESC Heart Fail. 2022 Dec;9(6):4198-4208. doi: 10.1002/ehf2.14154. Epub 2022 Sep 13. PMID 36101502
- [Derived] Tang Y, Yao L, Liu Z, Ma X, Luo Q, Zhao Z, Huang Z, Tu L, Gao L, Jin Q, Ni X, Xiong C. Effect of calcium channel blockers evaluated by cardiopulmonary exercise testing in idiopathic pulmonary arterial hypertension responding to acute pulmonary vasoreactivity testing. Pulm Pharmacol Ther. 2017 Apr;43:26-31. doi: 10.1016/j.pupt.2017.01.012. Epub 2017 Feb 1. PMID 28159512